CLINICAL TRIAL: NCT02370186
Title: The Role of Dysfunctional HDL in Severe Sepsis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UFJ 2014-193; IRB201702454 (Other: IRB-01)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Severe Sepsis; Septic Shock; Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe sepsis results in over 300,000 Emergency Department (ED) visits and 215,000 deaths annually in the US. Currently there are no effective drug therapies for sepsis. High density lipoprotein (HDL) has antioxidant, anti-inflammatory, and antithrombotic properties and is protective in sepsis. Its functions in sepsis are primarily mediated by its main apolipoprotein, Apo-A1, that: 1) neutralize potent bacterial toxins, 2) protect blood vessel walls from damage, 3) prevent tissue damage through antioxidant properties, and 4) mediate thymocyte apoptosis (critical for survival) and endogenous corticosteroid release. However, recent literature presents inconsistent data on HDL functionality and shows that HDL becomes non-functional during acute inflammatory states called dysfunctional HDL (Dys-HDL). Several causes for Dys-HDL have been hypothesized including the presence of Apo A1 polymorphisms, which may worsen the pathologic inflammatory response in sepsis and have been demonstrated in early sepsis, making Dys-HDL an unstudied potential early marker. This project aims to: 1) determine the presence of Dys-HDL in adult patients with early severe sepsis who present to the ED (Dys-HDL will be tested using a novel cell free assay and HDL Inflammatory Index will be measured), and 2) examine the relationship between Dys-HDL and cumulative organ dysfunction via Sequential Organ Failure Assessment (SOFA) score. Results of this study could establish Dys-HDL as an early disease marker for sepsis which is influential in the development of sepsis-induced organ dysfunction.

DETAILED DESCRIPTION:
Sepsis is a systemic inflammatory response to infection, which leads to acute organ dysfunction and shock. Current therapies are aimed at normalizing hemodynamic parameters during early sepsis resuscitation to reduce mortality. The investigators hypothesize that future strategies should be personalized, and should target the mediators of the septic response on an individual patient basis. One of these mediators is HDL which works by facilitating clearance of bacterial toxins, maintaining the integrity of the endothelium, and preventing inflammation, a function performed by Apo-A1. The association of HDL with cardiovascular health has been well-studied in the Caucasian and Asian populations, where research has demonstrated that HDL can become pro-inflammatory and thus may not perform its functions of being anti-inflammatory, anti-thrombotic and anti-oxidant. Such HDL is called Dys-HDL. Dys-HDL or pro-inflammatory HDL may play a pivotal role in sepsis, an area that has not been fully studied. The mechanism by which HDL becomes dysfunctional is one of debate, but the main hypothesis is through polymorphisms of Apo-A1, possibly via the myeloperoxidase enzyme, and each polymorphism produces different HDL levels and activity. These alterations can lead to increased susceptibility to septic death due to inability to neutralize lipopolysaccharide, loss of thymocyte apoptosis (critical for protection against sepsis) and endogenous corticosteroid release, and loss of the ability to preserve HDLs antioxidant properties. Dys-HDL has also been demonstrated in early sepsis and may serve as a potential early disease marker. For these reasons, the investigators believe that Dys-HDL may play a pivotal role in the sepsis cascade which leads to organ dysfunction and death. Aim 1. Determine the presence of Dys-HDL in adult patients with early severe sepsis who present to the ED. Aim 2. Examine the relationship between Dys-HDL and cumulative organ dysfunction as measured by the sequential organ failure assessment (SOFA) score, a validated measure of organ dysfunction in severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older with at least 2 of 4 SIRS criteria plus:

   * lactate ≥ 2 mg/dL, AND
   * SOFA Score ≥ 4* (see Appendix A), or

Exclusion Criteria:

* Patients <18 years of age
* Pregnant subjects
* No valid consent available
* Familial/genetic disorders of lipid metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who present to one Emergency Department and who meet criteria for severe sepsis or septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03-12 (Actual); Study Completion 2017-03-12 (Actual)

PRIMARY OUTCOMES:
Dys-HDL in adult patients with early severe sepsis | 48 hours
  Measure Dys-HDL in adult patients with early severe sepsis who present to the ED.

SECONDARY OUTCOMES:
Relationship between Dys-HDL and Cumulative Organ Dysfunction | 48 hours
  Examine the relationship between Dys-HDL and cumulative organ dysfunction as measured by the sequential organ failure assessment (SOFA) score.

CONTACTS AND LOCATIONS:
Overall Officials: Faheem W Guirgis, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guirgis FW, Dodani S, Leeuwenburgh C, Moldawer L, Bowman J, Kalynych C, Grijalva V, Reddy ST, Jones AE, Moore FA. HDL inflammatory index correlates with and predicts severity of organ failure in patients with sepsis and septic shock. PLoS One. 2018 Sep 14;13(9):e0203813. doi: 10.1371/journal.pone.0203813. eCollection 2018. PMID 30216360